CLINICAL TRIAL: NCT01002859
Title: Double-Blind Phase II Pilot Monocentric Randomized Clinical Trial Evaluating the Effect of a Preliminary Administration of Cyclosporine on Different Markers of Cardiac Ischemia Led by the Aortic Cross-clamp During Coronary Artery Bypass Surgery With Cardiopulmonary Bypass.
Brief Title: Effect of Preliminary Administration of Cyclosporine (Sandimmun ®) on Different Markers of Cardiac Ischaemia Induced by Cardiopulmonary Bypass
Acronym: Ciclo et CEC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulties to include patients
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DCIC 08 04
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Artery Bypass Surgery; Cardiopulmonary Bypass
Keywords: Coronary artery bypass graft surgery (CABG); Cardiopulmonary Bypass (CPB); Cyclosporine; ischaemia reperfusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cyclosporin (Active Comparator): Intravenous cyclosporin injection.
  Interventions: Drug: Sandimmum
- Pacebo (Placebo Comparator): Intravenous injection of NaCl solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sandimmum — Intravenous injection of cyclosporine
  Arms: cyclosporin
Drug: Placebo — Intravenous Injection of NaCl solution
  Arms: Pacebo

SUMMARY:
Observe the effect of preliminary cyclosporine administration on different markers of cardiac ischaemia led by the aortic cross-clamp during coronary artery bypass surgery with Cardiopulmonary bypass.

DETAILED DESCRIPTION:
The coronary artery bypass surgery, in spite of substantial improvements during the last years, is still associated to a post-operative mortality and morbidity: myocardial infarction, heart failure, cardiac arrhythmia, renal failure, Stroke.

These complications are often due to ischaemia - reperfusion injury event. Recent studies showed that in case of cellular stress (in particular during the reperfusion after ischaemia) a not specific pore, called Mitochondrial permeability transition Pore (MPTP), could be opened. That caused the loss of ion homeostasis, then cell death as well as by apoptosis as by necrosis.

Prevent the opening of this MPTP during the myocardial reperfusion after coronary bypass, for example, is an important objective to improve the cardioprotection.

The Cyclosporin A, prevents the MPTP from opening. Several studies have shown an cytoprotection led by cyclosporin A, after ischaemia reperfusion in several models as isolated rats heart, in vivo rats heart and ex vivo myocardial ( atrial ) human tissues.

Recently, a multicentric study performed in humans, during the acute phase of myocardial infarction, showed a reduction of infarct size by approximately 40% in the cyclosporine group compared to control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for a coronary artery bypass surgery
* Not urgent surgery
* Left ventricular ejection fraction (LVEF)> 40 %
* 18 years and older
* patient who have sign the informed consent form
* Affiliation to the French Social Security.

Exclusion Criteria:

* Beating heart surgery with or without Cardiopulmonary Bypass
* Patient receiving another surgical gesture combined to the CABG
* Myocardial infarction or vascular cerebral attack less than 30 days
* Previous History of cardiac surgery;
* Renal failure (creatinine > 200 µmol/l)
* Uncontrolled hypertension
* hyperkaliemy;
* hyperuricemy;
* Acute Coronary Syndrome
* Malignant tumor
* Unchecked infection
* Previous intravenous administration of Sandimmun ®;
* allergy to ciclosporin, ethyl alcohol, castor oil or nitrogen
* Pregnant Woman, parturient without contraception, or breast-feeding
* Age < 18 years
* Patient who have not signed the form of consent;
* Patient Under guardianship or being the object of a legal protective measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under curve and maximal blood level of both troponin-T and Creatine Kinase-MB after cardiopulmonary bypass | at anaesthesia (ti), at the end of the cardiopulmonary bypass (t0), and 6 h, 12 h, 24 h,48h and 72h after the end of the cardiopulmonary bypass.

SECONDARY OUTCOMES:
Area under curve and maximal blood level of S100β protein | at anaesthesia (ti), at the end of the cardiopulmonary bypass (t0), and 6 h, 12 h, 24 h,48h and 72h after the end of the cardiopulmonary bypass
Spontaneous defibrillation at aorta declamping; Post surgical atrial fibrillation; ECG (new Q wave); Transthoracic Echocardiogram (diastolic and systolic function study, research of paradoxical septal motion, study of cardiac output)....) | until Day 3 after the end of the cardiopulmonary bypass
Levels of inflammatory cytokines (TNF alpha , IL-1 alpha et IL-1 beta, IL-6, IL-8, IL-10). C-reactive protein (CRP) level | until day 8 after the end of the cardiopulmonary bypass
Creatine blood levels | until 3 months after the end of the cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Vincent BACH, MD, Principal Investigator — Cardiac Surgery Department - University Hospital of Grenoble,
Locations (1):
- Department of cardiac surgery - University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Crompton M. The mitochondrial permeability transition pore and its role in cell death. Biochem J. 1999 Jul 15;341 ( Pt 2)(Pt 2):233-49. PMID 10393078
- [Background] Halestrap AP, Clarke SJ, Javadov SA. Mitochondrial permeability transition pore opening during myocardial reperfusion--a target for cardioprotection. Cardiovasc Res. 2004 Feb 15;61(3):372-85. doi: 10.1016/S0008-6363(03)00533-9. PMID 14962470
- [Background] Hausenloy DJ, Duchen MR, Yellon DM. Inhibiting mitochondrial permeability transition pore opening at reperfusion protects against ischaemia-reperfusion injury. Cardiovasc Res. 2003 Dec 1;60(3):617-25. doi: 10.1016/j.cardiores.2003.09.025. PMID 14659807
- [Background] Shanmuganathan S, Hausenloy DJ, Duchen MR, Yellon DM. Mitochondrial permeability transition pore as a target for cardioprotection in the human heart. Am J Physiol Heart Circ Physiol. 2005 Jul;289(1):H237-42. doi: 10.1152/ajpheart.01192.2004. PMID 15961375
- [Background] Piot C, Croisille P, Staat P, Thibault H, Rioufol G, Mewton N, Elbelghiti R, Cung TT, Bonnefoy E, Angoulvant D, Macia C, Raczka F, Sportouch C, Gahide G, Finet G, Andre-Fouet X, Revel D, Kirkorian G, Monassier JP, Derumeaux G, Ovize M. Effect of cyclosporine on reperfusion injury in acute myocardial infarction. N Engl J Med. 2008 Jul 31;359(5):473-81. doi: 10.1056/NEJMoa071142. PMID 18669426